CLINICAL TRIAL: NCT04168853
Title: Cardiopulmonary Bypass and Internal Thoracic Arteries: Can Roller or Centrifugal Pumps Change Vascular Reactivity of the Grafts
Brief Title: Impact of Pumps on Internal Thoracic Arteries (IPITA)
Acronym: IPITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CHU Angers
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Coronary Disease
Keywords: cardiopulmonary bypass; pulsatility; systemic inflammatory response; arterial graft
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: The IPITA (Impact of Pumps on Internal Thoracic Arteries) study consisted of two parallel prospective, monocenter, randomized, active-treatment-controlled clinical trials
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roller pump group (Other): CABG was performed under normothermic (36-37°C) cardiopulmonary bypass (CPB). All components of the circuits were coated with phosphorylcholine inert surface (PHISIO, Sorin®). The pump manufacturer is Maquet® for the roller pumps.1.5 cm of ITA distality was sampled before blood flow interruption into the graft and before starting CPB (Time 1) and another segment (1.5 cm) before the last coronary anastomosis during aortic cross clamping (Time 2) (Figure 1). Each arterial segment was cut into three parts: a fresh part for arterial myography bathed and stored in a 50 ml organ bath containing a physiological salt solution (PSS). The other two parts were cooled in liquid nitrogen and stored at -80°C for immunohistochemistry and RT-PCR analysis.
  Interventions: Diagnostic Test: vascular reactivity of internal thoracic arteries
- Centrifugal pump group (Other): CABG was performed under normothermic (36-37°C) cardiopulmonary bypass (CPB). All components of the circuits were coated with phosphorylcholine inert surface (PHISIO, Sorin®). The pump manufacturer is Sorin® for the centrifugal pumps.1.5 cm of ITA distality was sampled before blood flow interruption into the graft and before starting CPB (Time 1) and another segment (1.5 cm) before the last coronary anastomosis during aortic cross clamping (Time 2) (Figure 1). Each arterial segment was cut into three parts: a fresh part for arterial myography bathed and stored in a 50 ml organ bath containing a physiological salt solution (PSS). The other two parts were cooled in liquid nitrogen and stored at -80°C for immunohistochemistry and RT-PCR analysis.
  Interventions: Diagnostic Test: vascular reactivity of internal thoracic arteries

INTERVENTIONS:
Diagnostic Test: vascular reactivity of internal thoracic arteries — 1. Internal thoracic arteries analysis Myography Superoxide detection and confocal microscopy Immunochemistry Quantitative real time transcription-polymerase chain reaction (RT-PCR) analysis
  2. Blood sampling and biochemical analysis

SUMMARY:
Cardiopulmonary bypass (CPB) induces a systemic inflammatory response and affects the organ vascular bed. Experimentally, the lack of pulsatility alters myogenic tone of resistance arteries and increases the parietal inflammatory response. The purpose of this study was to compare the vascular reactivity and the inflammatory response of the internal thoracic arteries (ITAs) between patients undergoing coronary artery bypass grafting (CABG) under CPB with a roller pump or with a centrifugal pump.

DETAILED DESCRIPTION:
Eighty elective male patients undergoing CABG were selected using one or two internal thoracic arteries under CPB with a roller pump (RP group) or centrifugal pump (CFP group). ITA samples were collected before starting CPB (Time 1) and before the last coronary anastomosis during aortic cross clamping (Time 2). Terminal complement complex activation (SC5b-9) and neutrophil activation (elastase) analysis were performed on arterial blood at the same times.

ELIGIBILITY:
Inclusion Criteria:

* male patients and elective coronary artery bypass grafting using at least one of the two ITAs.

Exclusion Criteria:

* female patients because their complement activation has been shown to be greater than that in men during surgery under cardiopulmonary bypass ; age < 18 years; CABG requiring additional valve repair or replacement; emergency surgery and insufficient length of the internal thoracic artery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Myography | 1 day
  for each patient, 2 fresh segments of ITA (Time 1 and Time 2) stored in PSS were analyzed. On day+1, these segments were mounted on a wire-myograph (DMT, Aarhens, DK) . Two tungsten wires (25 μm diameter) were inserted into the lumen of the arteries and connected to a force transducer and a micrometer, respectively. The arteries were bathed in the PSS solution. Wall tension, equivalent to intra-arterial pressure (90 mmHg), was applied and the blood vessels were allowed to stabilize for thirty minutes. Arterial contractility was assessed with phenylephrine (PE, 10 μmol/L). Acetylcholine-induced (Ach 10 μmol/L) relaxation was then obtained after phenylephrine-induced preconstruction (50% of maximal contraction) in the presence or in the absence of the NO synthesis blocker L-NMMA (3.10-4 mol/L) and in the presence or in the absence of the COX synthesis blocker Indomethacin (10-5 mol/L).

SECONDARY OUTCOMES:
Superoxide detection and confocal microscopy | 1 day
  : dihydroethidium staining (DHE, Sigma-Aldrich) was used to evaluate the in-situ levels of superoxide anions (O2-). DHE is permeable to cells and is oxidized by superoxide (O2-) to fluorescent products that are trapped by intercalation into the DNA. Sections (10 μm thickness) were incubated with DHE (1 μmol/L) in phosphate-buffered solution (PBS) and DAPI (4',6'-diamidino-2-phénulindole-Molecular probes, Invitrogen) for nuclear cells Fluorescent images of ethidium bromide were obtained using a confocal microscope (Nikon Eclipse TE2000S).
Immunochemistry | 1 day
  sections (10 μm thickness) of arteries were rehydrated by 500 μl of PBS during 10 minutes and fixated with 200 μl of paraformaldehyde (PFA) (pH = 7.4, room temperature) and then were rinsed by PBS. Permeabilization with 200 μl of PBS-BSA (Bovine Serum Albumin - Sigma) 10% - Tween 0.1% during 40 minutes and then saturation with PBS-BSA 10% during 40 minutes were performed. Sections were incubated overnight with 100 μl of anti-CD45 antibody at 1/500th dilution for leukocyte staining or anti-CD80 antibody at 1/200th dilution for lymphocyte staining. Antibodies were labelled with a red fluorochrome (Phycoerythrine). Karyoplasm was stained blue by DAPI solution. On day+1, sections were rinsed with PBS and analyzed with the confocal microscope. Fluorescent images were quantified with the ImageJ (NIH) software.
Quantitative real time transcription-polymerase chain reaction (RT-PCR) analysis | 1 day
  Sections of ITAs were dried and stored at -80°C in RNA later Stabilization Reagent (Qiagen). RNA extraction was performed using the RNeasy® micro kit (Qiagen). 500 ng of RNA extracted from each artery were used to synthesize cDNA using the QuantiTect® Reverse Transcription kit (Qiagen). Quantitative real-time PCR was performed with Sybr® Green PCR Master Mix (Applied Biosystems) using a Light cycler 480 Real-Time PCR System (Roche).
Blood sampling and biochemical analysis | 2 hours
  Serial arterial blood samples for elastase and for SC5b-9, marker of terminal complement complex activation, were collected at Time 1 and Time 2. Specimens were centrifuged (10 minutes, 3,000 rpm, 4°C) immediately to obtain plasma which was stored at - 80°C before analysis.
  Enzyme-linked immunosorbent assay techniques were used from 10 μl of plasma to measure terminal complement (SC5b-9; Quidel, San Diego, CA, USA) and 50 μl of plasma for neutrophil elastase (Neutrophil ELA2, Assay pro, St Charles, USA). The limit of sensitivity of each assay undertaken was as follows: SC5b-9 = 16 ng/mL and elastase = 20 ng/mL.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fouquet O, Dang Van S, Baudry A, Meisnerowski P, Robert P, Pinaud F, Binuani P, Chretien JM, Henrion D, Baufreton C, Loufrani L. Cardiopulmonary bypass and internal thoracic artery: Can roller or centrifugal pumps change vascular reactivity of the graft? The IPITA study: A randomized controlled clinical trial. PLoS One. 2020 Jul 9;15(7):e0235604. doi: 10.1371/journal.pone.0235604. eCollection 2020. PMID 32645079